CLINICAL TRIAL: NCT02760953
Title: A Multi Center, Randomized, Parallel Controlled Study of Applying Transurethral Resection of Bladder Tumor With Adjuvant Cryoablation to Treat Bladder Cancer
Brief Title: TURBt With Adjuvant Cryoablation to Treat Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Zhongshan Hospital (Other); Shanghai 5th People's Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Haowen Jiang, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENSCURE-2015-BCC
Record Dates: First submitted 2016-04-22; First posted 2016-05-04 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Bladder Cancer; Cryoablation
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cryosurgery; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUR with Cryoablation (Experimental): Patients received TUR to treat bladder cancer and immediate cryoablation was applied on the tumor bed in order to eliminate possible residual tumor. Two or three cycles of freeze could be give to fully cover the lesion. One cycle last three to five minutes base on our previous animal experiments.
  Interventions: Procedure: Cryoablation
- TUR with instant instillation (Active Comparator): Patients received TUR to treat bladder cancer and pirarubicin instillation was given within 24 hours after TUR. This is in accord with the current guideline.
  Interventions: Drug: Epirubicin

INTERVENTIONS:
Procedure: Cryoablation — Using a novel cryoablation unit to perform transurethral cryoablation on the tumor base after transurethral resection
  Arms: TUR with Cryoablation
Drug: Epirubicin — Epirubicin instillation should be give within 24 hours after initial TUR, this is accord with current guideline.
  Arms: TUR with instant instillation

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of applying cryoablation as an adjuvant therapy with TUR to treat bladder tumor.

DETAILED DESCRIPTION:
Bladder tumors are one of the most commonly diagnosed urinary tumors in the world. Worldwide, it has been estimated that 429,800 new cases of and 165,100 deaths due to bladder tumor occurred in 2012. Transurethral resection (TUR) is the gold-standard treatment for non-muscle invasive bladder cancer (NMIBC). In muscle-invasive bladder cancer, TUR also plays a vital role as a bladder-sparing procedure regardless of whether it is applied as a monotherapy or in combination with chemo-radiotherapy.

Whether radical resection of a tumor is initially performed can be essential in the treatment of bladder tumors. Incomplete TUR influences a patient's prognosis, regardless of whether it is part of a NMIBC treatment or part of bladder-sparing trimodal therapy. However, the quality of TUR is one of the greatest concerns in the treatment of bladder tumor. After initial TUR, approximately 70% of patients exhibit incomplete resection re-staging TUR. Of these patients, 30% exhibit residual tumors at the resection site. To solve this problem, a second TUR 4-6 weeks after the initial TUR is recommended by the guidelines, and these repeated TURs detect residual tumors in 26-83% of cases.

The investigators sought to identify other therapies that can be combined with TUR to eliminate residual tumors. As a minimally invasive method, cryotherapy has been widely used for urological tumors, including prostate tumor and kidney tumor. With respect to bladder tumors, cryotherapy remains in the exploration phase. Only a few studies of the use of computed tomography (CT)-guided percutaneous cryoablation for the treatment of bladder cancer have been reported. Unlike solid viscera, such as the prostate or kidney, the bladder exhibits the features of hollow viscera. Cryoablation through the transurethral approach could be possible if the safety of the procedure can be ensured. Our recent animal study conducted in a porcine model demonstrated the feasibility and safety of transurethral focal, full-thickness cryoablation. No perforations were observed during two eight-minute freeze cycles. Based on the success of transurethral cryoablation in animal experiments, the investigators performed this study to explore the safety and efficacy of cryoablation as an adjuvant therapy with TUR in the treatment of bladder tumors.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed bladder tumor, stage T1 or T2
* Number of lesions ≤ 3
* Tumor size ≤ 3cm

Exclusion Criteria:

* With other malignant diseases
* T3 or above
* Enlarged pelvic lymph node or distant metastasis
* Poor overall condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-19 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Residual tumor rate | 4-6 weeks after surgery
  The investigators would perform reTUR 4-6 weeks after initial surgery to detect residual tumor

SECONDARY OUTCOMES:
Indwelling time | One month after surgery
Adverse event rate | Through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Haowen Jiang, Doctor, Study Director — Huashan Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu S, Zou L, Mao S, Zhang L, Xu H, Yang T, Jiang H, Ding Q. The safety and efficacy of bladder cryoablation in a beagle model by using a novel balloon cryoprobe. Cryobiology. 2016 Apr;72(2):157-60. doi: 10.1016/j.cryobiol.2016.02.007. Epub 2016 Mar 3. PMID 26939677
- [Background] Hruby GW, Marruffo F, Ortiz J, Durak E, Edelstein A, Levi G, Landman J. Transurethral bladder cryoablation in the porcine model. Urology. 2007 Aug;70(2):391-5. doi: 10.1016/j.urology.2007.03.028. PMID 17826526
- [Derived] Xu C, Jiang S, Zou L, Sheng L, Shi G, Xu B, Wang Z, Xu D, Xie X, Luo J, Guo J, Jiang H. Endoscopic balloon cryoablation plus transurethral resection for bladder cancer: A phase 2, multicenter, randomized, controlled trial. Cancer. 2023 Feb 1;129(3):415-425. doi: 10.1002/cncr.34563. Epub 2022 Dec 7. PMID 36477612